CLINICAL TRIAL: NCT05722431
Title: Délibération éthique en réanimation, Impact de la Mise en Place de réunions éthiques formalisées, Une étude Pilote
Brief Title: Ethical Deliberation in the Intensive Care Unit, Impact of Formalized Multidisciplinary Team Meetings, a Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DER
Record Dates: First submitted 2023-01-11; First posted 2023-02-10 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Ethics, Narrative
Keywords: End of life decisions in the ICU; Multidisciplinary team meetings; Ethical decision making climate; Nurses job satisfaction
MeSH Terms: conditions — Narration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Most patients who die in the intensive care unit do so after a withholding or withdrawing of life sustaining treatments (WWLST) decision. The implementation of formalized interdisciplinary team meetings for ethical deliberation in the ICU may improve nurses participation in WWLST decisions. The investigators decided to implement such team meetings in their ICU. At this occasion, the investigators will measure job satisfaction, job related frustration and ethical decision making climate climate.

DETAILED DESCRIPTION:
Most patients who die in the intensive care unit do so after a withholding or withdrawing of life sustaining treatments (WWLST) decision. Because those decisions are value-laden, guidelines as well as french regulations recommend that they should involve not only medical doctors but also nurses. Despite that, nurses' involvement remains incomplete. Poor collaboration between doctors and nurses on ethical decisions is associated with job dissatisfaction, burnout and desire to quit. The implementation of formalized interdisciplinary team meetings for ethical deliberation in the ICU may improve nurses participation in WWLST decisions.

For those reasons the investigators decided to implement such team meetings in their ICU. At this occasion, the investigators will measure job satisfaction, job related frustration and ethical decision making climate climate.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted in the ICU

Exclusion Criteria:

* Age below 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in the ICU
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in nurses perception of ethical decision making climate in the ICU | june 2023, january 2024
  Nurses answers to the questionnaire "Ethical Decision-Making Climate Questionnaire (7 factors evaluated, for each factor score ranges from 1 to 5, higher scores indicate a better climate)".

SECONDARY OUTCOMES:
Change in nurses psychological well being at work | 2 evaluations: may 2023, january 2024
  Nurses answers to the Index of psychological well being at work (5 factors, for each factor score ranges from 1 to 5, higher scores indicate more well being).
Change in nurses frustration of job's related psychological needs | 2 evaluations: may 2023, january 2024
  Nurses answers to the Job related psychological needs frustration score (3 factors, for each factor score ranges from 1 to 5, higher score indicate more frustration)
Change in nurses desire to leave | 2 evaluations: may 2023, january 2024
  Nurses answers to a one question questionnaire:
  "I have thoughts about leaving my current position/job" (lickert scale, score range from 1 to 5, higher score indicate a higher desire to leave)
Non beneficial care | January 2024
  Duration of mechanical ventilation in patients who ultimately die (number of days)

CONTACTS AND LOCATIONS:
Overall Officials: ROMAIN MIGUEL MONTANES, MD, Principal Investigator — University Hospital of TOURS; Servane Barrault, PhD, Principal Investigator — University of Tours
Locations (1):
- Trauma and surgical intensive care unit, Tours University Hospital, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided